CLINICAL TRIAL: NCT00750997
Title: Hypertonic Modulation of Inflammation Following Injury
Status: Terminated | Type: Observational
Why Stopped: Enrollment in the clinical trial was stopped for futility
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Eileen Bulger, Professor, Surgery, University of Washington
Other Study IDs: 28233
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Hemorrhagic Shock; Traumatic Brain Injury
MeSH Terms: conditions — Shock, Hemorrhagic; Brain Injuries, Traumatic | interventions — Saline Solution, Hypertonic; Dextrans

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hypertonic saline: Hypertonic resuscitation
  Interventions: Drug: hypertonic saline
- Control: normal saline: Normal saline resuscitation

INTERVENTIONS:
Drug: hypertonic saline — patients in parent trial were randomized to 250cc 7.5% saline, 7.5%saline with 6%dextran or normal saline as control as the initial resuscitation fluid after injury with signs of either hemorrhagic shock or severe traumatic brain injury
  Other Names: hypertonic saline with dextran
  Groups: Hypertonic saline

SUMMARY:
This project seeks to determine the effect of prehospital resuscitation with hypertonic saline vs. conventional crystalloids on the inflammatory response after injury. The leading cause of late mortality following injury is multiple organ dysfunction syndrome (MODS), which results from a dysfunctional inflammatory response after injury. Previous studies suggest that hypertonic saline may be beneficial by modulating this initial response and decreasing subsequent organ injury. This project takes advantage of a unique opportunity, afforded by an NIH-funded multi-center clinical trial of hypertonic resuscitation (conducted by the Resuscitation Outcomes Consortium), to obtain blood samples from patients enrolled in this trial to analyze inflammatory responses early after hypertonic vs. conventional resuscitation. This study was an ancillary study to the main randomized clinical trial and thus prospective observational in nature

The proposed study will be carried out in experiments grouped in three Specific Aims: Aim 1 provides a thorough investigation of the immunomodulatory response following hypertonic resuscitation with regard to neutrophil, monocyte, and T cell responses at serial time points after injury and resuscitation. Aim 2 comprises experiments to investigate the mechanisms by which hypertonicity may alter inflammatory cell signaling. Aim 3 seeks to correlate the laboratory findings with clinical endpoints reflective of immune dysfunction including inflammation, organ failure, nosocomial infection, and sepsis.

The investigators hypothesize that hypertonic resuscitation will be associated with modulation of the excessive inflammatory response seen after injury and thus will result in reduced rates of inflammatory organ injury.

DETAILED DESCRIPTION:
This was an ancillary study to the larger clinical trials of prehospital hypertonic resuscitation conducted by the resuscitation outcomes consortium. This study investigated markers of immune function and coagulation in a subset of patients enrolled in the larger trials at two of the clinical sites. Four publications detail the results please see references

ELIGIBILITY:
Inclusion Criteria:

* Blunt or Penetrating trauma with prehospital systolic blood pressure < 70 or 70-90 mmHg with Heart rate > 108 OR Blunt trauma with prehospital Glasgow coma score <= 8

Exclusion Criteria:

* Age < 15 yrs
* Known prisoners
* Pregnancy
* Ongoing Cardiopulmonary resuscitation (CPR)
* Burns < 20%
* Hypothermia < 28 C
* > 2 liters intravenous fluid prior to study fluid administration
* > 4 hour from time of dispatch

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled in clinical trial of Hypertonic Resuscitation based on prehospital evidence of hypovolemic shock or severe brain injury
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
neutrophil activation | Emergency department admission
  several parameters of neutrophil activation were assessed

SECONDARY OUTCOMES:
Endothelial cell activation | Emergency department admission
  several parameters of endothelial cell activation were assessed
coagulation parameters | Emergency department admission
  several parameters of coagulation were assessed
monocyte activation | Emergency department admission
  several parameters of monocyte activation were assessed

CONTACTS AND LOCATIONS:
Overall Officials: Eileen M Bulger, MD, Principal Investigator — University of Washington
Locations (2):
- University of Washington, Seattle, Washington, United States
- University of Toronto, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No
Data from the primary RCT will be made available through the Resuscitation Outcomes consortium. This was an ancillary study

REFERENCES:
- [Result] Delano MJ, Rizoli SB, Rhind SG, Cuschieri J, Junger W, Baker AJ, Dubick MA, Hoyt DB, Bulger EM. Prehospital Resuscitation of Traumatic Hemorrhagic Shock with Hypertonic Solutions Worsens Hypocoagulation and Hyperfibrinolysis. Shock. 2015 Jul;44(1):25-31. doi: 10.1097/SHK.0000000000000368. PMID 25784523
- [Result] Junger WG, Rhind SG, Rizoli SB, Cuschieri J, Baker AJ, Shek PN, Hoyt DB, Bulger EM. Prehospital hypertonic saline resuscitation attenuates the activation and promotes apoptosis of neutrophils in patients with severe traumatic brain injury. Shock. 2013 Nov;40(5):366-74. doi: 10.1097/SHK.0000000000000038. PMID 24088993
- [Result] Junger WG, Rhind SG, Rizoli SB, Cuschieri J, Shiu MY, Baker AJ, Li L, Shek PN, Hoyt DB, Bulger EM. Resuscitation of traumatic hemorrhagic shock patients with hypertonic saline-without dextran-inhibits neutrophil and endothelial cell activation. Shock. 2012 Oct;38(4):341-50. doi: 10.1097/SHK.0b013e3182635aca. PMID 22777113
- [Result] Bulger EM, Tower CM, Warner KJ, Garland T, Cuschieri J, Rizoli S, Rhind S, Junger WG. Increased neutrophil adenosine a3 receptor expression is associated with hemorrhagic shock and injury severity in trauma patients. Shock. 2011 Nov;36(5):435-9. doi: 10.1097/SHK.0b013e318231ee2e. PMID 21841534